CLINICAL TRIAL: NCT00762372
Title: Phase 2/3 Clinical Study With BLM-240 in Adult Surgery Patients That Need General Anesthesia
Brief Title: Japan Phase 2/3 Clinical Study With BLM-240 (Desflurane)
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Baxter Healthcare Corporation (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: BLM-240-003
Record Dates: First submitted 2008-09-26; First posted 2008-09-30 (Estimated); Results first posted 2019-03-08 (Actual); Last update posted 2019-03-08 (Actual); Status verified 2018-11

CONDITIONS: Anesthesia
Keywords: anesthesia; desflurane
MeSH Terms: interventions — Desflurane; Nitrous Oxide; Sevoflurane

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- desflurane (Experimental)
  Interventions: Drug: desflurane
- desflurane/N2O (Experimental)
  Interventions: Drug: desflurane/nitrous oxide
- sevoflurane/N2O (Active Comparator)
  Interventions: Drug: sevoflurane/nitrous oxide

INTERVENTIONS:
Drug: desflurane — volatile liquid for inhalation
  Other Names: Suprane; BLM-240
  Arms: desflurane
Drug: desflurane/nitrous oxide — volatile liquid for inhalation with gas for inhalation
  Other Names: Suprane; BLM-240; N2O
  Arms: desflurane/N2O
Drug: sevoflurane/nitrous oxide — volatile liquid for inhalation and gas for inhalation
  Other Names: sevoflurane; N2O
  Arms: sevoflurane/N2O

SUMMARY:
The purposes of this study are to evaluate the efficacy and safety of desflurane (BLM-240) as an anesthetic agent and to demonstrate the non-inferiority of desflurane to sevoflurane in term of awakening/recovery from anesthesia.

DETAILED DESCRIPTION:
The study evaluates the efficacy and safety of the use of desflurane (BLM-240) (with and without nitrous oxide) in maintenance of general anesthesia in adult patients undergoing surgical procedures typically performed under general anesthesia in Japan (thoracic, abdominal, joints, back, and neck), where analgesics and muscle relaxants are concomitantly used. The study is also intended to demonstrate the non-inferiority of desflurane with nitrous oxide to sevoflurane with nitrous oxide in time to awakening/recovery.

ELIGIBILITY:
Inclusion Criteria:

* ASA PS 1-3
* age: older than 19 y and younger than 70 y
* undergoing surgery of the thorax(thoracotomy, thoracotomy plus laparotomy, endoscopy; but excluding cardiovascular),abdomen(laparotomy,endoscopy;but excluding cesarean section), joints (including peripheral vessels), back (spine)or neck (neck, throat)
* willing to be hospitalized for at least 3 days and 2 nights (from the day before surgery to the day after surgery)
* having given written consent

Exclusion Criteria:

* need for spinal subarachnoid, epidural or local anesthesia (except local surface or infiltration anesthesia for catheter insertion or use of local anesthetic for testing before inserting epidural catheter for post-surgical pain)
* contraindication for use of nitrous during surgery
* anticipated need for postoperative transfer to intensive care unit and receive mechanical pulmonary ventilation
* BMI of 30 kg/m2 or more
* serious hepatic, renal, or circulatory disorder (Grade 3 per Notification 80 by MHW, Pharmaceutical Affairs Bureau, Safety Division)
* uncontrollable hypertension (SBP 160 mmHg or higher while on antihypertensive therapy)
* emergency surgery
* history of hypersensitivity to components of sevoflurane, fentanyl, propofol, vecuronium or other anesthetic
* contraindication to sevoflurane, fentanyl, propofol, or vecuronium
* exposure or suspected exposure to inhalational halogenated anesthetic within 3 mo prior to consent
* known or suspected history or family history of malignant hyperthermia
* considered likely to have difficulty in receiving tracheal intubation due to conditions such as brachygnathia, micrognathia, bucked teeth, articular rheumatism or injury of cervical spine/cervical cord
* known or suspected to be pregnant or lactating
* participated in a clinical study within 6 mo prior to consent
* history of drug dependence
* history of epilepsy
* otherwise judged by the investigator to be unsuitable for the study

Ages: 20 Years to 69 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 216 (Actual)
Dates: Start 2008-02; Primary Completion 2008-08 (Actual); Study Completion 2008-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Junzo Takeda, MD, Principal Investigator — School of Medicine, Keio University
Locations (15):
- Japan (15):
  - Kagoshima University Medical and Dental University, Kagoshima
  - Kyoto University, Kyoto
  - Nagoya University, Nagoya
  - Okayama University, Okayama
  - Osaka University, Osaka
  - Sapporo Medical University, Sapporo
  - Hamamatsu University, Shizuoka
  - Jikei University, Tokyo
  - Juntendo University, Tokyo
  - Keio University, Tokyo
  - Nippon Medical School, Tokyo
  - NTT East Japan Kanto Medical, Tokyo
  - Tokai University, Tokyo
  - Tokyo University, Tokyo
  - Tokyo Women's Medical University, Tokyo

RESULTS

PARTICIPANT FLOW:
Groups:
- BLM 240 N2O Group: Inhalation of BLM-240 was initiated at 3% (vaporizer dial setting) with N2O at 50-70%. The inspired concentration was adjusted depending on the patient's condition during anesthetic maintenance (gas flow rate: 2 to 6 L/min).
- BLM 240 O2 Group: Inhalation of BLM-240 was initiated at 3% (vaporizer dial setting) with o2 (>=30%). The inspired concentration was adjusted depending on the patient's condition during anesthetic maintenance (gas flow rate: 2 to 6 L/min).
- Sevoflurane Group: Inhalation of sevoflurane was initiated at 1% (vaporizer dial setting) with N2O at 50-70%. The inspired concentration was adjusted depending on the patient's condition during anesthetic maintenance (gas flow rate: 2 to 6 L/min).
Period: Overall Study
Arm/Group | BLM 240 N2O Group | BLM 240 O2 Group | Sevoflurane Group
Started | 111 (N=114 enrolled but 3 participant's discontinued before start of study drug administration.) | 55 (N=57 enrolled but 2 participant's discontinued before start of study drug administration.) | 50 (N=53 enrolled but 3 participant's discontinued before start of study drug administration.)
Completed | 110 | 55 | 50
Not Completed | 1 | 0 | 0
Not completed — Adverse Event | 1 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | BLM 240 N2O Group | BLM 240 O2 Group | Sevoflurane Group | Total
Number analyzed (Participants) | 111 | 55 | 50 | 216
Age, Continuous [Mean (Standard Deviation); unit: years] | 48.5 (12.2) | 47.4 (13.6) | 45.7 (13.4) | 47.2 (11.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 60 | 35 | 31 | 126
  Male | 51 | 20 | 19 | 90
Race/Ethnicity, Customized [Number; unit: participants]
  Japan | 111 | 55 | 50 | 216

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Body Movement During Anesthetic Maintenance
Description: The investigator or sub-investigator observed the patient for body movement (excluding bucking) during anesthetic maintenance.
Time Frame: Day 1 (During surgery, duration ranging <2 hours, 2-4 hours, and ≥4 hours)
Population: Full Analysis Set (FAS) - subjects assigned to treatment groups, excluding subjects with significant GCP violations (significant violations regarding informed consent and study procedures), subjects who did not receive the allocated study drug, subjects whose ASA status was not Class I, II, III, or subjects for whom no data were available.
Measure: Number; unit: participants
Groups:
- BLM-240 Group: Cumulative summary of two BLM 240 treatment Arms, including N2O and O2.
- BLM-240 N2O Group: Inhalation of BLM-240 was initiated at 3% (vaporizer dial setting) with N2O at 50-70%. The inspired concentration was adjusted depending on the patient's condition during anesthetic maintenance (gas flow rate: 2 to 6 L/min).
- BLM-240 O2 Group: Inhalation of BLM-240 was initiated at 3% (vaporizer dial setting) with o2 (>=30%). The inspired concentration was adjusted depending on the patient's condition during anesthetic maintenance (gas flow rate: 2 to 6 L/min).
Arm/Group | BLM-240 Group | BLM-240 N2O Group | BLM-240 O2 Group | Sevoflurane Group
Number analyzed (Participants) | 166 | 111 | 55 | 50
participants
  No | 165 | 111 | 54 | 50
  Yes | 1 | 0 | 1 | 0

2. Primary Outcome: Number of Participants With Recall/Memory Issues During Anesthetic Maintenance
Description: The investigator or sub-investigator observed the patient for the presence or absence of awakening during anesthetic maintenance and interviewed the patient on the day after surgery to confirm whether the patient has any memory during anesthetic maintenance.
Time Frame: Day 1 (During surgery, duration ranging <2 hours, 2-4 hours, and ≥4 hours)
Population: FAS
Measure: Number; unit: participants
Arm/Group | BLM-240 Group | BLM-240 N2O Group | BLM-240 O2 Group | Sevoflurane Group
Number analyzed (Participants) | 166 | 111 | 55 | 50
participants
  No | 165 | 110 | 55 | 50
  Yes | 0 | 0 | 0 | 0
  Unevaluable | 1 | 1 | 0 | 0

3. Primary Outcome: Number of Participants Requiring Rescue Treatment During Anesthetic Maintenance
Description: Rescue medication includes vasopressors and depressors.
Time Frame: Day 1 (During surgery, duration ranging <2 hours, 2-4 hours, and ≥4 hours)
Population: FAS
Measure: Number; unit: participants
Arm/Group | BLM-240 Group | BLM-240 N2O Group | BLM-240 O2 Group | Sevoflurane Group
Number analyzed (Participants) | 166 | 111 | 55 | 50
participants
  No | 120 | 75 | 45 | 34
  Yes | 46 | 36 | 10 | 16

4. Primary Outcome: Number of Participants Not Receiving Rescue Treatment Whose Blood Pressure/Heart Rate Maintained Above/Below 70%
Description: "Rescue medication includes vasopressors and depressors. Percentage of observation points at which systolic pressure 80 to <150 mmHg and heart rate 50 to <100 bpm could be maintained "
Time Frame: Day 1 (During surgery, duration ranging <2 hours, 2-4 hours, and ≥4 hours)
Population: FAS
Measure: Number; unit: participants
Arm/Group | BLM-240 Group | BLM-240 N2O Group | BLM-240 O2 Group | Sevoflurane Group
Number analyzed (Participants) | 166 | 111 | 55 | 50
participants
  >=70% | 111 | 68 | 43 | 31
  <70% | 9 | 7 | 2 | 3

5. Primary Outcome: Number of Participants Receiving Rescue Treatment Whose Blood Pressure/Heart Rate Maintained Above/Below 70%
Description: Rescue medication includes vasopressors and depressors. Percentage of observation points at which no rescue treatment was judged to be required based on blood pressure/heart rate
Time Frame: Day 1 (During surgery, duration ranging <2 hours, 2-4 hours, and ≥4 hours)
Population: FAS
Measure: Number; unit: participants
Arm/Group | BLM-240 Group | BLM-240 N2O Group | BLM-240 O2 Group | Sevoflurane Group
Number analyzed (Participants) | 166 | 111 | 55 | 50
participants
  >=70% | 46 | 36 | 10 | 16
  <70% | 0 | 0 | 0 | 0

6. Primary Outcome: Overall Assessment of Efficacy
Description: Evaluation on the efficacy (ability) of BLM-240 as an anesthetic drug.
Time Frame: Day 1 (During surgery, duration ranging <2 hours, 2-4 hours, and ≥4 hours)
Population: FAS
Measure: Number; unit: participants
Arm/Group | BLM-240 Group | BLM-240 N2O Group | BLM-240 O2 Group | Sevoflurane Group
Number analyzed (Participants) | 166 | 111 | 55 | 50
participants
  Excellent Ability | 111 | 68 | 43 | 31
  Sufficient Ability | 9 | 7 | 2 | 3
  Some Ability | 44 | 35 | 9 | 16
  Insufficient Ability | 1 | 0 | 1 | 0
  Inadequate | 0 | 0 | 0 | 0
  Unevaluable | 1 | 1 | 0 | 0

7. Primary Outcome: Time to Extubation
Description: Evaluation of Awakening/Recovery from Anesthesia from end of study drug inhalation to extubation. The patient was extubated when the following signs were observed:(1) clear consciousness, (2) ability to breathe spontaneously (minute ventilation >=50 mL/kg/min), and (3) stable circulatory dynamics (systolic pressure: >=100 mmHg).
Time Frame: Day 1 (Post-Surgery, from end of study drug inhalation to extubation)
Population: FAS
Measure: Mean (Standard Deviation); unit: minutes
Arm/Group | BLM-240 Group | BLM-240 N2O Group | BLM-240 O2 Group | Sevoflurane Group
Number analyzed (Participants) | 166 | 111 | 55 | 50
minutes | 9.8 (5) | 10.1 (4.6) | 9.3 (5.7) | 14.8 (8.4)
Statistical Analysis 1: Comparison: BLM-240 N2O Group vs Sevoflurane Group; Test type: Non-Inferiority — Time to extubation = treatment group + surgical site +surgery time; Mean Difference (Final Values) = -4.6, 95% CI 2-sided [-6.6 to -2.7], Standard Error of Mean 1.0

8. Secondary Outcome: Time to Awakening
Description: Time from the end of study drug inhalation. After the end of inhalation of the study drug, the investigator commanded the patient to open his/her eyes once every minute to check whether he/she awoke and recorded the time of awakening.
Time Frame: Day 1 (Post-Surgery, from the end of study drug inhalation to awakening)
Population: FAS
Measure: Mean (Standard Deviation); unit: minutes
Arm/Group | BLM-240 Group | BLM-240 N2O Group | BLM-240 O2 Group | Sevoflurane Group
Number analyzed (Participants) | 166 | 111 | 55 | 50
minutes | 6.8 (4) | 7.2 (3.7) | 6.2 (4.6) | 10.4 (5.5)
Statistical Analysis 1: Comparison: BLM-240 N2O Group vs BLM-240 O2 Group; Test type: Non-Inferiority — Adjusted means of "time from the end of study drug inhalation to extubation" in the BLM-240 N2O group and sevoflurane group, which were obtained by analysis of covariance with surgical site and surgery time as covariates, were used to verify the non-inferiority of BLM-240 to the comparator sevoflurane, with a delta = 1.0 (minute) and significance level alpha = 2.5% (one-sided); p = 0.1500, t-test, 2 sided

9. Secondary Outcome: Time to Stating Birth Date
Description: After extubation, the investigator called and asked the patient to state the birth date once every minute and recorded the time the patient could state the birth date. Time from the end of study drug inhalation.
Time Frame: Day 1 (Post-Surgery, after extubation)
Population: FAS
Measure: Mean (Standard Deviation); unit: minutes
Arm/Group | BLM-240 Group | BLM-240 N2O Group | BLM-240 O2 Group | Sevoflurane Group
Number analyzed (Participants) | 166 | 111 | 55 | 50
minutes | 11.4 (5.4) | 11.8 (5.3) | 10.6 (5.6) | 16.2 (8.7)
Statistical Analysis 1: Comparison: BLM-240 N2O Group vs BLM-240 O2 Group; Test type: Non-Inferiority — Two-sample t-test; p = 0.0001, t-test, 2 sided

10. Secondary Outcome: Time to Reaching an Aldrete Score >=8 (Min)
Description: Score includes a ranking of 0-2 (higher shows improvement) in activity, respiration, circulation, consciousness, and O2 saturation (SpO2). After extubation, the investigator observed the patient's condition every 5 minutes until the Aldrete score reached >=8 and recorded the Aldrete scores at 5-minute intervals.
Time Frame: Day 1 (Post-Surgery, after extubation)
Population: FAS
Measure: Mean (Standard Deviation); unit: minutes
Arm/Group | BLM-240 Group | BLM-240 N2O Group | BLM-240 O2 Group | Sevoflurane Group
Number analyzed (Participants) | 166 | 111 | 55 | 50
minutes | 13.6 (5.2) | 13.9 (4.8) | 13.1 (6) | 18.7 (8.4)

11. Secondary Outcome: Time to Clear Consciousness
Description: "Clear consciousness" means that patients responded to investigator's command for physical movement such as "hold my finger tight."
Time Frame: Day 1 (Post-Surgery, from awakening to before extubation)
Population: FAS
Measure: Mean (Standard Deviation); unit: minutes
Arm/Group | BLM-240 Group | BLM-240 N2O Group | BLM-240 O2 Group | Sevoflurane Group
Number analyzed (Participants) | 166 | 111 | 55 | 50
minutes | 7.7 (4.4) | 8.1 (4.2) | 6.9 (4.7) | 12.3 (7.4)

12. Secondary Outcome: Changes in Bispectral Index (BIS) Over Time During Anethetic Maintenance
Description: BIS is used to monitor depth of anesthesia. The BIS monitor provides a single number, which ranges from 0 (equivalent to EEG silence) to 100. A BIS value between 40 and 60 generally indicates an appropriate level for general anesthesia.
Time Frame: Day 1 (During surgery, duration ranging <2 hours, 2-4 hours, and ≥4 hours)
Population: FAS
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | BLM-240 N2O Group | BLM-240 O2 Group | Sevoflurane Group
Number analyzed (Participants) | 111 | 55 | 50
score on a scale
  Prior to start of inhalation | 50.7 (13.2) | 48.6 (14.8) | 49.8 (12.6)
  End of inhalation | 46.3 (12.9) | 57.3 (18.6) | 48.8 (11.8)
  After Awakening | 84.8 (15.4) | 88.2 (10.8) | 87.4 (11.2)
  Before Extubation | 90.1 (11.9) | 90.8 (10.8) | 90.9 (9.9)
  5 minutes after extubation | 93.5 (6.7) | 95.2 (5.3) | 93.4 (6.1)

13. Secondary Outcome: Number of Participants Requiring Rescue Medication Due to Rise in Blood Pressure or Heart Rate
Description: Rescue medication can include vasopressors and depressors.
Time Frame: Day 1 (During surgery, duration ranging <2 hours, 2-4 hours, and ≥4 hours)
Population: FAS
Measure: Number; unit: participants
Arm/Group | BLM-240 Group | BLM-240 N2O Group | BLM-240 O2 Group | Sevoflurane Group
Number analyzed (Participants) | 166 | 111 | 55 | 50
participants | 6 | 4 | 2 | 0
Statistical Analysis 1: Comparison: BLM-240 N2O Group vs Sevoflurane Group; Test type: Non-Inferiority — Fisher's exact test; p = 0.3113, Fisher Exact

14. Secondary Outcome: Number of Participants Requiring Rescue Medication Due to Drop in Blood Pressure or Heart Rate
Description: Rescue medication can include vasopressors and depressors.
Time Frame: Day 1 (During surgery, duration ranging <2 hours, 2-4 hours, and ≥4 hours)
Population: FAS
Measure: Number; unit: participants
Arm/Group | BLM-240 Group | BLM-240 N2O Group | BLM-240 O2 Group | Sevoflurane Group
Number analyzed (Participants) | 166 | 111 | 55 | 50
participants | 40 | 32 | 8 | 16

15. Secondary Outcome: Number of Participants Requiring Rescue Medication Due to Arrhythmia
Description: Rescue medication can include vasopressors and depressors.
Time Frame: Day 1 (During surgery, duration ranging <2 hours, 2-4 hours, and ≥4 hours)
Population: FAS
Measure: Number; unit: participants
Arm/Group | BLM-240 Group | BLM-240 N2O Group | BLM-240 O2 Group | Sevoflurane Group
Number analyzed (Participants) | 166 | 111 | 55 | 50
participants | 3 | 1 | 2 | 0
Statistical Analysis 1: Comparison: BLM-240 N2O Group vs Sevoflurane Group; Test type: Non-Inferiority — Fisher's exact test; p = 1.0000, Fisher Exact

16. Secondary Outcome: Range of End-Tidal Anesthetic Percent Concentrations During Anesthetic Maintenance
Description: Measurement by infrared absorption spectrometry. The concentrations of BLM-240 and sevoflurane at the start of inhalation were set at 3% and 1%,respectively (by vaporizer dial setting). Concentrations are monitored to determine which levels keep the patient in stable condition without requiring rescue treatment.
Time Frame: Day 1 [just before the start of inhalation of study drug, during anesthetic maintenance (every 5 minutes after the start of inhalation of study drug), at the end of inhalation of study drug, immediately after awakening, and just before extubation]
Population: FAS
Measure: Number; unit: percentage
Arm/Group | BLM-240 N2O Group | BLM-240 O2 Group | Sevoflurane Group
Number analyzed (Participants) | 111 | 55 | 50
percentage
  Low Range | 3 | 4 | 1.2
  High Range | 4 | 5 | 1.4

17. Secondary Outcome: Range of Inspired Anesthetic Concentrations Below End-Tidal Anesthetic Percent Concentrations During Anesthetic Maintenance
Description: Measurement by infrared absorption spectrometry. Ranges reflecting when concentrations were stable. The inspired concentration was adjusted depending on the patient's condition during anesthetic maintenance (gas flow rate: 2 to 6 L/min).
Time Frame: Day 1 [just before the start of inhalation of study drug, during anesthetic maintenance (every 5 minutes after the start of inhalation of study drug), at the end of inhalation of study drug, and just before extubation]
Population: FAS
Measure: Number; unit: percentage
Arm/Group | BLM-240 Group | Sevoflurane Group
Number analyzed (Participants) | 166 | 60
percentage
  Low Range | 0.3 | 0.1
  High Range | 0.5 | 0.3

18. Secondary Outcome: End-Tidal Anesthetic Percent Concentrations Successfully Maintained Anesthesia
Description: Successfully maintaining anesthesia is defined as keeping the patient in stable condition (systolic pressure 80 to <150 mmHg and heart rate 50 to <100bpm) without requiring rescue treatment or additional dose of opioid analgesics (<=2 ug/kg/hr).If patient was found to have body movement, recall, or memory during anesthetic maintenance, data for such patient were to be excluded from summary statistic calculation.
Time Frame: as for outcome 16
Population: FAS
Measure: Mean (Standard Deviation); unit: percentage
Arm/Group | BLM-240 Group | BLM-240 N2O Group | BLM-240 O2 Group | Sevoflurane Group
Number analyzed (Participants) | 166 | 111 | 55 | 50
percentage | 3.97 (1.17) | 3.69 (1.06) | 4.48 (1.21) | 1.30 (0.39)

ADVERSE EVENTS:
Time Frame: 3 Days before study drug through 7 days after surgery.
Arm/Group | BLM 240 Group | BLM 240 N2O Group | BLM 240 O2 Group | Sevoflurane Group
All-Cause Mortality (participants affected / at risk) | 0/166 | 0/111 | 0/55 | 0/50
Serious Adverse Events (participants affected / at risk) | 0/166 | 5/111 | 0/55 | 2/50
Other Adverse Events (participants affected / at risk) | 163/166 | 108/111 | 55/55 | 49/50
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | BLM 240 Group (N=166) | BLM 240 N2O Group (N=111) | BLM 240 O2 Group (N=55) | Sevoflurane Group (N=50)
Altered state of consciousness (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Respiratory arrest (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Suture rupture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pyelonephritis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Cardiac arrest (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Loss of consciousness (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pneumonia (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Haematocrit decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Haemoglobin decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | BLM 240 Group (N=166) | BLM 240 N2O Group (N=111) | BLM 240 O2 Group (N=55) | Sevoflurane Group (N=50)
Anaemia (Blood and lymphatic system disorders) | 2 (2) | 1 (1) | 1 (1) | 2 (2)
Arrhythmia supraventricular (Cardiac disorders) | 2 (2) | 1 (1) | 1 (1) | 0 (0)
Atrioventricular block complete (Cardiac disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Bundle branch block (Cardiac disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Cardiac arrest (Cardiac disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Nodal rhythm (Cardiac disorders) | 2 (2) | 2 (2) | 0 (0) | 0 (0)
Sinus arrhythmia (Cardiac disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Sinus tachycardia (Cardiac disorders) | 1 (1) | 1 (1) | 0 (0) | 1 (1)
Supraventricular extrasystoles (Cardiac disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Tachycardia (Cardiac disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Ventricular extrasystoles (Cardiac disorders) | 3 (3) | 2 (2) | 1 (1) | 0 (0)
Tinnitus (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Vitreous floaters (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Conjunctival hyperaemia (Eye disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Abdominal distension (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 3 (3) | 2 (2) | 1 (1) | 0 (0)
Abdominal pain lower (Gastrointestinal disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Abdominal pain upper (Gastrointestinal disorders) | 2 (2) | 0 (0) | 2 (2) | 1 (1)
Abdominal tenderness (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Ascites (Gastrointestinal disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Constipation (Gastrointestinal disorders) | 17 (17) | 12 (12) | 5 (5) | 8 (8)
Diarrhoea (Gastrointestinal disorders) | 4 (4) | 3 (3) | 1 (1) | 1 (1)
Dysphagia (Gastrointestinal disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Faeces discoloured (Gastrointestinal disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Lip swelling (Gastrointestinal disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Nausea (Gastrointestinal disorders) | 55 (55) | 38 (38) | 17 (17) | 8 (8)
Stomach discomfort (Gastrointestinal disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Stomatitis (Gastrointestinal disorders) | 2 (2) | 1 (1) | 1 (1) | 1 (1)
Swollen tongue (Gastrointestinal disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Vomiting (Gastrointestinal disorders) | 28 (29) | 20 (21) | 8 (8) | 5 (5)
Anal inflammation (Gastrointestinal disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Gastrointestinal motility disorder (Gastrointestinal disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Chills (General disorders) | 5 (5) | 4 (4) | 1 (1) | 1 (1)
Feeling abnormal (General disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Feeling hot (General disorders) | 1 (1) | 0 (0) | 1 (1) | 1 (1)
Granuloma (General disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Local swelling (General disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Oedema peripheral (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pain (General disorders) | 26 (27) | 16 (17) | 10 (10) | 10 (10)
Peripheral coldness (General disorders) | 1 (1) | 1 (1) | 0 (0) | 1 (1)
Pyrexia (General disorders) | 45 (45) | 27 (27) | 18 (18) | 12 (12)
Swelling (General disorders) | 5 (5) | 3 (3) | 2 (2) | 2 (2)
Infusion site swelling (General disorders) | 1 (1) | 0 (0) | 1 (1) | 1 (1)
Nasopharyngitis (Infections and infestations) | 2 (2) | 2 (2) | 0 (0) | 0 (0)
Pneumonia (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pyelonephritis (Infections and infestations) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Wound infection (Infections and infestations) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Joint dislocation (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Tooth injury (Injury, poisoning and procedural complications) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
XIth nerve injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Suture rupture (Injury, poisoning and procedural complications) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Mouth injury (Injury, poisoning and procedural complications) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Contusion (Injury, poisoning and procedural complications) | 1 (1) | 1 (1) | 0 (0) | 1 (1)
Wound complication (Injury, poisoning and procedural complications) | 106 (108) | 73 (75) | 33 (33) | 28 (29)
Post procedural haematoma (Injury, poisoning and procedural complications) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Alanine aminotransferase increased (Investigations) | 14 (14) | 9 (9) | 5 (5) | 2 (2)
Aspartate aminotransferase increased (Investigations) | 15 (15) | 11 (11) | 4 (4) | 3 (3)
Blood amylase increased (Investigations) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Blood bilirubin increased (Investigations) | 27 (27) | 14 (14) | 13 (13) | 4 (4)
Blood chloride decreased (Investigations) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Blood cholesterol increased (Investigations) | 3 (3) | 2 (2) | 1 (1) | 0 (0)
Blood creatinine increased (Investigations) | 2 (2) | 2 (2) | 0 (0) | 0 (0)
Blood lactate dehydrogenase increased (Investigations) | 12 (12) | 8 (8) | 4 (4) | 3 (3)
Blood potassium decreased (Investigations) | 7 (7) | 4 (4) | 3 (3) | 1 (1)
Blood potassium increased (Investigations) | 5 (5) | 3 (3) | 2 (2) | 1 (1)
Blood pressure decreased (Investigations) | 18 (21) | 13 (16) | 5 (5) | 10 (12)
Blood pressure increased (Investigations) | 5 (7) | 2 (4) | 3 (3) | 0 (0)
Blood sodium decreased (Investigations) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Blood triglycerides increased (Investigations) | 18 (18) | 13 (13) | 5 (5) | 8 (8)
Blood urea increased (Investigations) | 2 (2) | 1 (1) | 1 (1) | 0 (0)
Blood uric acid decreased (Investigations) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Blood uric acid increased (Investigations) | 2 (2) | 2 (2) | 0 (0) | 1 (1)
Body temperature decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Body temperature increased (Investigations) | 2 (2) | 2 (2) | 0 (0) | 1 (2)
C-reactive protein increased (Investigations) | 3 (3) | 2 (2) | 1 (1) | 0 (0)
Electrocardiogram ST segment depression (Investigations) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Gamma-glutamyltransferase increased (Investigations) | 23 (23) | 16 (16) | 7 (7) | 4 (4)
Glucose urine present (Investigations) | 17 (17) | 15 (15) | 2 (2) | 3 (3)
Haematocrit decreased (Investigations) | 11 (11) | 7 (7) | 4 (4) | 1 (1)
Haematocrit increased (Investigations) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Blood urine present (Investigations) | 53 (53) | 36 (36) | 17 (17) | 19 (19)
Haemoglobin decreased (Investigations) | 11 (11) | 7 (7) | 4 (4) | 1 (1)
Haemoglobin increased (Investigations) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Heart rate decreased (Investigations) | 15 (15) | 14 (14) | 1 (1) | 7 (7)
Heart rate increased (Investigations) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Oxygen saturation decreased (Investigations) | 4 (4) | 3 (3) | 1 (1) | 0 (0)
Platelet count decreased (Investigations) | 2 (2) | 1 (1) | 1 (1) | 1 (1)
Red blood cell count decreased (Investigations) | 12 (12) | 8 (8) | 4 (4) | 1 (1)
Red blood cell count increased (Investigations) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Respiratory rate decreased (Investigations) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Volume blood decreased (Investigations) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
White blood cell count decreased (Investigations) | 3 (3) | 1 (1) | 2 (2) | 0 (0)
White blood cell count increased (Investigations) | 57 (57) | 43 (43) | 14 (14) | 17 (17)
Platelet count increased (Investigations) | 15 (15) | 10 (10) | 5 (5) | 5 (5)
Protein urine present (Investigations) | 17 (17) | 12 (12) | 5 (5) | 1 (1)
Blood alkaline phosphatase increased (Investigations) | 7 (7) | 5 (5) | 2 (2) | 1 (1)
Urine output decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Anorexia (Metabolism and nutrition disorders) | 2 (2) | 1 (1) | 1 (1) | 0 (0)
Fluid retention (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Gout (Metabolism and nutrition disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Hypocalcaemia (Metabolism and nutrition disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Tetany (Metabolism and nutrition disorders) | 1 (1) | 1 (1) | 0 (0) | 1 (1)
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1) | 0 (0) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 7 (7) | 4 (4) | 3 (3) | 3 (3)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 1 (1) | 2 (3)
Myalgia (Musculoskeletal and connective tissue disorders) | 2 (2) | 1 (1) | 1 (1) | 0 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Musculoskeletal stiffness (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Altered state of consciousness (Nervous system disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Epilepsy (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Facial palsy (Nervous system disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Headache (Nervous system disorders) | 18 (18) | 9 (9) | 9 (9) | 7 (7)
Hypoaesthesia (Nervous system disorders) | 6 (6) | 5 (5) | 1 (1) | 1 (1)
Loss of consciousness (Nervous system disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Somnolence (Nervous system disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Insomnia (Psychiatric disorders) | 15 (15) | 9 (9) | 6 (6) | 7 (7)
Restlessness (Psychiatric disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Bladder pain (Renal and urinary disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Dysuria (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Urethral pain (Renal and urinary disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1) | 0 (0) | 2 (2)
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 7 (7) | 5 (5) | 2 (2) | 0 (0)
Foreign body aspiration (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Laryngeal oedema (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Nasal congestion (Reproductive system and breast disorders) | 2 (2) | 1 (1) | 1 (1) | 0 (0)
Pharyngeal oedema (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Pharyngolaryngeal pain (Respiratory, thoracic and mediastinal disorders) | 9 (9) | 6 (6) | 3 (3) | 7 (7)
Productive cough (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 1 (1) | 1 (1) | 0 (0)
Respiratory arrest (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 2 (2) | 0 (0) | 0 (0)
Respiratory depression (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Wheezing (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Sputum retention (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 1 (1) | 1 (1)
Pharyngolaryngeal discomfort (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 2 (2) | 0 (0) | 0 (0)
Blister (Skin and subcutaneous tissue disorders) | 3 (3) | 2 (2) | 1 (1) | 0 (0)
Decubitus ulcer (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Dermatitis contact (Skin and subcutaneous tissue disorders) | 5 (5) | 2 (2) | 3 (3) | 3 (3)
Eczema (Skin and subcutaneous tissue disorders) | 2 (2) | 1 (1) | 1 (1) | 0 (0)
Erythema (Skin and subcutaneous tissue disorders) | 5 (5) | 3 (3) | 2 (2) | 3 (3)
Haemorrhage subcutaneous (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Pruritus (Skin and subcutaneous tissue disorders) | 2 (2) | 2 (2) | 0 (0) | 1 (1)
Rash (Skin and subcutaneous tissue disorders) | 3 (3) | 1 (1) | 2 (2) | 0 (0)
Skin exfoliation (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Urticaria (Skin and subcutaneous tissue disorders) | 4 (4) | 2 (2) | 2 (2) | 0 (0)
Hypertension (Vascular disorders) | 2 (2) | 1 (1) | 1 (1) | 0 (0)
Orthostatic hypotension (Vascular disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Wound haemorrhage (Vascular disorders) | 3 (3) | 2 (2) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes